CLINICAL TRIAL: NCT05900557
Title: Neurologic Deficits and Recovery in Chronic Subdural Hematoma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI has left the institution
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1454683
Record Dates: First submitted 2023-05-18; First posted 2023-06-12 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Chronic Subdural Hematoma
MeSH Terms: conditions — Hematoma, Subdural, Chronic

STUDY DESIGN:
Intervention Model Description: Single arm study performing subdural ECoG monitoring to assess for presence or absence of spreading depolarization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ECoG monitoring (Experimental): Patients undergoing standard of care surgical evacuation of cSDH. will have subdural ECoG monitoring electrode placed crossing frontal and temporal lobes for 1-5 days of post operative monitoring. All subjects will undergo long term followup testing.
  Interventions: Diagnostic Test: ECoG monitoring

INTERVENTIONS:
Diagnostic Test: ECoG monitoring — Brief (1-5 days) of post operative ECoG monitoring to detect spreading depolarization.

SUMMARY:
Chronic subdural hematoma (cSDH) is one of the most common problems treated by neurosurgeons, particularly as the population ages. While often dismissed as a benign problem, it has become clear that cSDH is associated with worse long term functional and cognitive outcomes compared to matched controls. Though surgical techniques for treatment of cSDH are becoming more effective and safe, a persisting problem of fluctuating, stroke-like neurological deficits has re-emerged. Such deficits are not always directly related to hematoma mass effect and not always relieved with surgical decompression, but can result in prolonged hospital course, additional workup, and sometimes even additional invasive treatments. While the cause of such events is unknown, we recently documented for the first time that massive waves of spreading depolarization can occur in these patients and were closely linked to such neurologic deficits in some patients. In the current study, we plan to expand on these preliminary findings with rigorous, standardized application of post operative subdural electrocorticography monitoring, pioneered at our institution to detect SD. We also plan to build on our large retrospective analysis estimating the overall incidence of such deficits in cSDH patients by assessing multiple proposed risk factors for SD. In addition, for the first time, we will assess the short- and long-term consequences of cSDH and SD with detailed functional, cognitive, and headache related outcome measurement. These assessments are based on several remarkable cases we have observed with time-locked neurologic deterioration associated with recurrent SD. This study qualifies as a mechanistic clinical trial in that we will be prospectively assigning patients to the intervention of SD monitoring and assessing outcomes related to the occurrence of SD. This constitutes the application of a novel measure of brain signaling and assessing biomarkers of these physiologic processes of SD. These studies will provide critically needed information on this novel mechanism for neurologic deficits and worse outcomes after cSDH evacuation. Upon successful completion, we would identify a targetable mechanism for poor outcomes that occur commonly in patients with cSDH. This overall strategy offers the opportunity to radically improve the care of patients with cSDH by focusing on clinical trials of pharmacologic therapies for neurologic deficits in patients with cSDH.

ELIGIBILITY:
Inclusion Criteria:

* chronic/ subacute subdural hematoma deemed necessary for surgical evacuation,
* Ability to consent or have LAR consent

Exclusion Criteria:

* emergent need for evacuation,
* acute traumatic subdural hematoma, and
* severe baseline disability (mRS>2) (modified Rankin Scale)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Post operative neurologic deterioration. | 1-5 days
  Incidence of decline in Markwalder grading scale (0[normal]-4[comatose]) or Glasgow coma scale (3[no response] to 15[normal]) by one point.

SECONDARY OUTCOMES:
eGOS | 30day, 90 day, 180 day
  Extended Glasgow outcome scale 1(dead)- 8(upper good recovery)
MoCA | 30day, 90 day, 180 day
  Montreal Cognitive Assessment (1-30) 30 is the best
NIH toolbox cognitive battery | 30day, 90 day, 180 day
  The NIH Toolbox Cognitive Battery provides an overall summary score along with fluid and crystallized cognition summary scores.
PROMIS 29 profile | 30day, 90 day, 180 day
  The PROMIS-29 v2.0 profile assesses pain intensity using a single 0-10 numeric rating item and seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance) using four items per domain
TBI QOL | 30day, 90 day, 180 day
  The TBI-QOL consists of 20 independent calibrated item banks and 2 uncalibrated scales that measure physical, emotional, cognitive, and social aspects of health-related quality of life
Headache disability Index | 30day, 90 day, 180 day
  The Headache Disability Index (HDI) is a 27-item questionnaire.The first two questions asks the patient to identify the frequency (1 per month; more than 1 but less than 4 per month; more than 1 per week) and intensity (mild, moderate, severe) of their headache. The remaining questions evaluate quality of life issues to determine headache disability.

IPD SHARING:
Plan to Share IPD: No